CLINICAL TRIAL: NCT04535180
Title: Sarcopenia and Osteoporosis in the Patients With Hemophilia
Status: Completed | Type: Observational
Sponsor: Tri-Service General Hospital (Other)
Responsible Party: Principal Investigator, Tsung-Ying Li, Attending physician, Tri-Service General Hospital
Other Study IDs: 1-107-05-053
Record Dates: First submitted 2020-08-12; First posted 2020-09-01 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Sarcopenia; Hemophilia; Osteoporosis, Osteopenia; Hemophilic Arthropathy
MeSH Terms: conditions — Sarcopenia; Hemophilia A; Osteoporosis; Bone Diseases, Metabolic | interventions — Absorptiometry, Photon

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemophilia
  Interventions: Diagnostic Test: Dual-energy X-ray absorptiometry (DXA)

INTERVENTIONS:
Diagnostic Test: Dual-energy X-ray absorptiometry (DXA) — Body composition will be measured using whole-body DXA (GE Lunar iDXA, GE Healthcare Lunar, Madison, Wisconsin, U.S.A.). Extremity skeletal muscle mass will be calculated using the values measured via the DXA; ASM will be calculated as the sum of skeletal muscle mass in the arms and legs, assuming that the mass of lean soft tissue is a skeletal muscle. Appendicular skeletal mass index (ASM/Ht2 ) will be determined as the sum of the arm and leg lean mass (kg)/height2 (m2
  ). BMD will be measured in lumbar spine and bilateral hip by the same DXA device (GE Lunar iDXA, GE Healthcare Lunar, Madison, Wisconsin, U.S.A.)

SUMMARY:
Hemophilia is a bleeding disorder and repeated joint bleeding leads to hemophilic arthropathy. Among patients with hemophilia, vitamin D deficiency and hemophilic arthropathy have been associated with osteoporosis in several clinical studies.There is no data on the prevalence of osteoporosis in hemophilia patients in Taiwan or Asia. To the best of our knowledge, no previous studies have reported the prevalence of sarcopenia and correlation with osteoporosis in hemophilia adult patients. This study will investigate the prevalence and corelation of sarcopenia and low BMD in patients with hemophilia.

patients in Taiwan. The study will estimate the prevalence of sarcopenia and body composition in the hemophilia population and compared baseline demographic and clinical characteristics between the non-sarcopenia and sarcopenia individuals, with particular emphasis on the overlap with osteoporosis and hemophilic arthropathy.

ELIGIBILITY:
Inclusion Criteria:

* Hemophilia patients

Exclusion Criteria:

* History of total hip arthroplasty
* History of instrumentation in lumbar spine

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hemophilia adult patients
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Sacropenia | up to 4 weeks
  Extremity skeletal muscle mass will be calculated using the values measured via the DXA

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided